CLINICAL TRIAL: NCT05878613
Title: Effect of Treadmill Training With and Without Trunk Kinesiotaping on Balance and Gait in Chronic Stroke Patients
Brief Title: Treadmill Training With Kinesiotaping Affects Balance and Gait in Chronic Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0206
Record Dates: First submitted 2023-04-18; First posted 2023-05-26 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Stroke
Keywords: balance; gait; kinesiotape; stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treadmill training with KT group (TTKT group) (Experimental): Participants will undergo treadmill training with kinesiotape applied on their trunk muscles/
  Interventions: Device: treadmill training with KT group (TTKT group)
- treadmill training without KT group (TT group) (Active Comparator): Participants will undergo treadmill training.
  Interventions: Device: treadmill training without KT group (TT group)

INTERVENTIONS:
Device: treadmill training with KT group (TTKT group) — The area to be taped will be cleaned with an alcohol swab, and the I-shaped elastic KT was applied to the four trunk muscles from their insertion to their origin. Patients will then undergo treadmill walking with easy speed control for 20 minutes. The training will be immediately stopped if the subject complain of fatigue during treadmill training; training will be resumed after sufficient rest.
  Arms: treadmill training with KT group (TTKT group)
Device: treadmill training without KT group (TT group) — General treadmill training without taping will be carried out for the same time as the gait training of the experimental group, and the treadmill speed will also be a comfortable speed in the same manner as in the experimental group.
  Arms: treadmill training without KT group (TT group)

SUMMARY:
The goal of this clinical trial is to determine the effects of treadmill training with and without trunk kinesiotaping on balance and gait of chronic stroke patients. The main question it aims to answer is:- Does kinesiotaping have added benefit to improve gait and balance in chronic stroke patients?.

Researcher will compare the treadmill training group with the group receiving treadmill training with kinesiotaping to see if there is any difference in the outcomes.

DETAILED DESCRIPTION:
Summary Stroke, one of the leading cause of death and disability worldwide, is defined as rapid deterioration of brain function due to disturbance in blood supply to the brain. According to the cause it is divided into two main types; ischemic stroke and hemorrhagic stroke. Stroke can lead to a number of physical impairments like muscle imbalance, impaired balance and postural control, poor voluntary control, body malalignment and disturbance of walking patterns etc. Ability to walk safely and participate in activities of daily living is the main goal of many individuals affected by stroke. Therefore, improving balance and gait is the primary focus of physical therapy interventions. Many therapeutic interventions such as , treadmill training, over ground gait training , Functional electrical stimulation, neurofacilitation approaches and strength training are used for improving balance and gait in patients affected by stroke, all of which have been proven to be beneficial. This study will be conducted to compare the effect of treadmill training with and without kinesiotaping on trunk muscles (rectus abdominis, erector spinae, external oblique and internal oblique) on gait and balance in chronic stroke patients.

Many studies have shown that trunk muscles have a very important role in balance and gait in patients with stroke and KT application may be an effective intervention for trunk function and postural control however, there is no evidence on whether providing support to the trunk with kinesiotaping during treadmill training will have any added benefit on balance and gait or not.

ELIGIBILITY:
Inclusion Criteria:

* both male and females
* Age 30-50 years.
* duration of onset of stroke >6 months.

Exclusion Criteria:

* • patients with orthopedic diseases(such as contracture) in the trunk and both lower extremities

  * A history of other neurologic diseases or disorders (MS, Parkinsons).
  * History of fall in last 6 months.'
  * History of unstable CVS diseases
  * high skin sensitivity or skin diseases
  * lower extremity surgery or fracture, low back pain, or allergy to the KT.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Berg Balance Scale (BBS): | 4th week
  The Berg Balance Scale (BBS) is a functional outcome measure in the International Classification of Functioning domain of activity, is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks. The BBS measures balance and functional mobility and has excellent reliability (0.99) and Interclass correlation coefficient 0.99 (0.98-0.99) .Berg balance scale scoring ranges from 0 to 56. The lower your score, the more at risk you are for losing your balance. In general, Berg balance scale scores are interpreted as such:
  0 to 20: A person with a score in this range will likely need the assistance of a wheelchair to move around safely.
  21 to 40: A person with a score in this range will need some type of walking assistance, such as a cane or a walker.
  41 to 56: A person with a score in this range is considered independent and should be able to move around safely without assistance.
  Changes from the baseline to 4th week
Dynamic gait index(DGI): | 4th week
  The DGI tests the ability of the participant to maintain walking balance while responding to different task demands, through various dynamic conditions. It is a useful test in individuals with vestibular and balance problems.Each item is scored on a scale of 0 to 3, with 3 indicating normal performance and 0 representing severe impairment. The best possible score on the DGI is a 24.A score of less than 19 indicates a risk for falling.
  total duration of intervention is 4 weeks (baseline measurement will be taken on week 1 and postinterventional measurement will be taken on week 4)

CONTACTS AND LOCATIONS:
Overall Officials: Wajiha Shahid, PhD, Principal Investigator — Riphah International University
Locations (1):
- Pakistan society of rehabilitation for disabled (PSRD), Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee YJ, Kim JY, Kim SY, Kim KH. The effects of trunk kinesio taping on balance ability and gait function in stroke patients. J Phys Ther Sci. 2016 Aug;28(8):2385-8. doi: 10.1589/jpts.28.2385. Epub 2016 Aug 31. PMID 27630439
- [Background] Rupasinghe CD, Ammar Bokhari S, Lutfi I, Noureen M, Islam F, Khan M, Amin F, Muthanna FMS. Frequency of Stroke and Factors Associated With It Among Old Age Hypertensive Patients in Karachi, Pakistan: A Cross-Sectional Study. Cureus. 2022 Mar 13;14(3):e23123. doi: 10.7759/cureus.23123. eCollection 2022 Mar. PMID 35425677
- [Background] Tally Z, Boetefuer L, Kauk C, Perez G, Schrand L, Hoder J. The efficacy of treadmill training on balance dysfunction in individuals with chronic stroke: a systematic review. Top Stroke Rehabil. 2017 Oct;24(7):539-546. doi: 10.1080/10749357.2017.1345445. Epub 2017 Jul 7. PMID 28687056
- [Background] Cho HY, Kim JS, Lee GC. Effects of motor imagery training on balance and gait abilities in post-stroke patients: a randomized controlled trial. Clin Rehabil. 2013 Aug;27(8):675-80. doi: 10.1177/0269215512464702. Epub 2012 Nov 5. PMID 23129815
- [Background] Hendrickson J, Patterson KK, Inness EL, McIlroy WE, Mansfield A. Relationship between asymmetry of quiet standing balance control and walking post-stroke. Gait Posture. 2014 Jan;39(1):177-81. doi: 10.1016/j.gaitpost.2013.06.022. Epub 2013 Jul 19. PMID 23877032
- [Background] Aprile I, Conte C, Cruciani A, Pecchioli C, Castelli L, Insalaco S, Germanotta M, Iacovelli C. Efficacy of Robot-Assisted Gait Training Combined with Robotic Balance Training in Subacute Stroke Patients: A Randomized Clinical Trial. J Clin Med. 2022 Aug 31;11(17):5162. doi: 10.3390/jcm11175162. PMID 36079092
- [Background] Beyaert C, Vasa R, Frykberg GE. Gait post-stroke: Pathophysiology and rehabilitation strategies. Neurophysiol Clin. 2015 Nov;45(4-5):335-55. doi: 10.1016/j.neucli.2015.09.005. Epub 2015 Nov 4. PMID 26547547
- [Background] Kim BR, Kang TW. The effects of proprioceptive neuromuscular facilitation lower-leg taping and treadmill training on mobility in patients with stroke. Int J Rehabil Res. 2018 Dec;41(4):343-348. doi: 10.1097/MRR.0000000000000309. PMID 30067555
- [Background] Kim WI, Choi YK, Lee JH, Park YH. The effect of muscle facilitation using kinesio taping on walking and balance of stroke patients. J Phys Ther Sci. 2014 Nov;26(11):1831-4. doi: 10.1589/jpts.26.1831. Epub 2014 Nov 13. PMID 25435710
- [Background] Dai S, Piscicelli C, Clarac E, Baciu M, Hommel M, Perennou D. Balance, Lateropulsion, and Gait Disorders in Subacute Stroke. Neurology. 2021 Apr 27;96(17):e2147-e2159. doi: 10.1212/WNL.0000000000011152. Epub 2020 Nov 11. PMID 33177223